CLINICAL TRIAL: NCT02932774
Title: Randomized, Double Blind, Parallel Group, Placebo Controlled, Multi-Center Study of the Efficacy and Safety of Zyrtec® (Cetirizine HCl) Syrup vs. Claritin® (Loratadine) Syrup vs. Placebo in Treatment of Children With Seasonal Allergic Rhinitis (SAR)
Brief Title: Randomized, Double Blind, Parallel Group, Placebo Controlled, Multi-Center Study of the Efficacy and Safety of Cetirizine HCl Syrup vs. Loratadine Syrup vs. Placebo in Treatment of Children With Seasonal Allergic Rhinitis (SAR)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A1431009
Record Dates: First submitted 2016-09-30; First posted 2016-10-13 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Allergic Rhinitis; Hay Fever; SAR; Rhinitis, Allergic, Seasonal
Keywords: SAR; seasonal allergic rhinitis; hay fever; seasonal allergic rhinoconjunctivitis
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis, Allergic, Seasonal | interventions — Cetirizine; Loratadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cetirizine 10 mg (Experimental): Cetirizine HCl 10 mg (1 mg/ml) syrup once daily for 2 weeks. Subjects who were randomized to receive cetirizine HCl syrup also received placebo syrup. Each subject was instructed to take 2 teaspoons from Bottle A and 2 teaspoons from Bottle B once daily, before 10:00 AM.
  Interventions: Drug: Cetirizine
- loratadine 10 mg (Active Comparator): Loratadine 10 mg (1 mg/ml) syrup once daily for 2 weeks. Subjects who were randomized to receive loratadine syrup also received placebo syrup. Each subject was instructed to take 2 teaspoons from Bottle A and 2 teaspoons from Bottle B once daily, before 10:00 AM.
  Interventions: Drug: Loratadine
- placebo (Placebo Comparator): Placebo syrup once daily for 2 weeks. Both placebo syrups were received by subjects who were randomized to receive placebo. Each subject was instructed to take 2 teaspoons from Bottle A and 2 teaspoons from Bottle B once daily, before 10:00 AM.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cetirizine — Cetirizine HCl 10 mg (1 mg/ml) syrup once daily before 10:00 AM for 2 weeks
  Other Names: ZYRTEC
  Arms: Cetirizine 10 mg
Drug: Loratadine — Loratadine HCl 10 mg (1 mg/ml) syrup once daily before 10:00 AM for 2 weeks
  Other Names: CLARITIN
  Arms: loratadine 10 mg
Other: Placebo — Placebo syrup once daily before 10:00 AM for 2 weeks
  Arms: placebo

SUMMARY:
The objective of this clinical trial was to assess the efficacy and safety of cetirizine HCl syrup vs. loratadine syrup vs. placebo syrup in the treatment of SAR in children 6 to 11 years old.

DETAILED DESCRIPTION:
This was a multi-center, randomized, double-blind, parallel-group, placebo-controlled, double dummy study of children with SAR conducted during the Spring tree and grass allergy season. Subjects qualified for randomization if the diary cards included (1) symptom scores of ≥2 for at least 2 of the following 4 rhinoconjunctivitis symptoms on 4 or more days: sneezing, runny nose, itchy eyes, and watery eyes; and (2) a total rhinoconjunctivitis (or Total Symptom Severity Complex [TSSC]) score of ≥5 on any 4 days. The TSSC score was expressed as the sum of the 4 individual symptoms scores recorded in the daily diary cards for the following symptoms: sneezing, runny nose, itchy eyes, and watery eyes.

Subjects were randomized to receive 1 of 3 treatments in a double-blind fashion using a 1:1:1 allocation ratio: cetirizine HCl syrup and placebo loratadine syrup; loratadine syrup and placebo cetirizine HCl syrup; or cetirizine placebo syrup and loratadine placebo syrup.

Number of Subjects (Planned and Analyzed): 1100 planned; 1536 screened; 683 randomized: 231 (33.8%) randomized to the cetirizine HCl treatment group, 221 (32.4%) to the loratadine treatment group, and 231 (33.8%) to the placebo treatment group.

Test Product and Reference Therapy: Subjects randomized to receive cetirizine HCl syrup also received placebo syrup; subjects randomized to receive loratadine syrup also received placebo syrup; and both placebo syrups were received by subjects randomized to receive placebo.

Duration of Double-Blind Treatment: 2 weeks.

Safety measures included the incidence and severity of treatment-emergent adverse events (AEs), vital signs, concomitant medications, and physical examination findings. Clinical laboratory evaluation was not required for this study.

Statistical Methods: All statistical tests related to treatment effect were 2-sided, and statistical significance was declared at the 0.05 probability level. Least squares means (LSMeans) were used to estimate treatment effect. Populations analyzed included the Full Analysis (intent-to-treat [ITT]) Set (FAS), Per-Protocol Set (PPS), Safety-Analyzable Set, and All-Screened Analysis Set. Demographic and baseline data for all subjects in the Safety-Analyzable Set were summarized and listed. The effects of treatment at the Overall and all other analysis Time Points were assessed using ANCOVA models. The main effects model contained terms for treatment and Investigator site, with baseline TSSC value as a covariate. The LSMeans and standard errors were based on the main effects model. Methods of analysis of secondary efficacy data included analysis of covariance (ANCOVA) models and Cochran-Mantel-Haenszel (CMH) row mean scores tests. Analysis of drug safety included the incidence of treatment-emergent AEs (TEAE), concomitant medications, vital signs, and physical examination findings for the Safety-Analyzable Set.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 6 to 11 years of age.
* Females who reached menarche either before or during the study, agreed to use acceptable methods of birth control if they became sexually active. Acceptable birth control was defined as oral contraceptives or Norplant®.
* Outpatient.
* History and diagnosis of seasonal allergic rhinitis (SAR) to a prevalent allergen (grass or tree).
* SAR to a prevalent allergen (grass or tree) of such severity that it required pharmacologic therapy each year for the last 2 consecutive years (including the present year).
* Documented SAR to a prevalent allergen (grass or tree) as confirmed by a recognized skin test (prick, intradermal [ID], or Multitest®) within the previous 15 months (Prick/Puncture wheal® ≥3 mm over the negative control; ID [up to concentration of 1:1000 w/v or 1000 protein nitrogen units (PNU)] wheal® ≥5 mm over the negative control). Documentation of SAR must have occurred at Visit 1 or within 15 months prior to Visit 1. If not performed at Visit 1, SAR testing must have been performed in the Principal Investigator's office or full documentation must have been available prior to randomization.
* Diary-recorded rhinoconjunctivitis symptom scores (24 hour reflective) that included at least two symptoms (sneezing, runny nose, itchy eyes, or watery eyes) at moderate severity (i.e., symptom score ≥2) on at least 4 days between Visits 1 and 2.
* Diary-recorded TSSC score ≥5 (based on the four symptoms noted in the criteria above) on any 4 days between Visits 1 and 2.
* Someone (subject and parent/legal guardian) from whom the Principal Investigator or study personnel would have expected conscientious cooperation over the duration of the study.
* A written informed assent must have been provided by the subject and a written informed consent must have been provided by the parent/legal guardian at Visit 1.

Exclusion Criteria:

* Had clinically significant nasal anatomical deformities with > 50% obstruction (i.e., septal defects, polyps).
* Experienced an episode of acute sinusitis or an upper respiratory tract infection (URTI) including otitis media and the common cold) within 21 days of Visit 1.
* Had a history of chronic sinusitis.
* Initiated or advanced an immunotherapy regimen during the course of the study. Subjects receiving a maintenance dose of immunotherapy were eligible.
* Had a history of attention deficit/hyperactivity disorder (ADHD) that was considered unstable by the Investigator, or if pharmacotherapy (i.e., Ritalin®, Adderall®) was required, subject must have been on pharmacotherapy for at least 1 month prior to Visit 1. The pharmacotherapeutic regimen was to remain stable during the conduct of the study.
* Had a history of learning disabilities or intellectual impairment that, in the opinion of the Investigator, would prevent the subject from participating in the study.
* Had impaired hepatic function (cirrhosis, hepatitis), glaucoma, or any symptomatic infection, any clinically significant hematologic, renal, endocrine, or gastrointestinal disease, and/or current neuropsychiatric condition with or without drug therapy, that was judged by the Investigator to be clinically significant and/or affect the subject's ability to participate in the clinical trial.
* Had a history of malignancy (except basal cell carcinoma), epilepsy or seizures (excluding febrile seizures), excessive alcohol intake or drug addiction, hypertension, or other clinically significant cardiovascular disease.
* Had a physical examination abnormality considered by the Investigator to be clinically significant and limiting to the study's conduct, unless the abnormality was related to underlying allergic rhinitis.
* Had a history of an allergy or hypersensitivity to cetirizine, loratadine, hydroxyzine, or any of their ingredients.
* Had asthma, which required any of the following within the past 30 days: 1) admission to the hospital, 2) emergency room visit, or 3) a change in dosing regimen. Subjects were allowed to continue theophylline, long acting β2 agonists, inhaled cromoglycate no more than 6.4 mg/day, or nedocrimil no more than 14 mg/day. Subjects were allowed to continue inhaled corticosteroids in doses not exceeding those listed in Appendix B of the study protocol, as long as the dose did not change during the study. Subjects were allowed the use of short acting β2 agonists on an as needed (PRN) basis.
* Had used intranasal or intra ophthalmic corticosteroids; oral leukotriene modifiers or leukotriene receptor antagonists within 14 days; or systemic (intramuscular and/or intravenous and/or oral) corticosteroids within 35 days prior to Visit 2. Topical corticosteroids for skin were allowed if covering ≤10% of body surface without occlusion.
* Used intranasal cromolyn (Nasalcrom®), optical cromolyn (Crolom®), ipratropium bromide (Atrovent® Nasal Spray), azelastine hydrochloride (Astelin® Nasal Spray), monamine oxidase (MAO) inhibitors, or beta blockers for the treatment of migraine headaches within 14 days prior to Visit 2.
* Used antiallergic ophthalmic treatments such as Acular®, Patanol®, or Alomide® within 7 days prior to Visit 2.
* Used H1-receptor antagonists (oral and topical), H2-receptor antagonists, or decongestants after Visit 1.
* Used tricyclic antidepressants, tranquilizers, or antiemetics of the phenothiazine class within 14 days prior to Visit 2.
* Used oral macrolide antibiotics or oral antifungals within 7 days prior to Visit 2.
* Used saline nasal spray or ocular drops (unless for contact lens use) within 72 hours prior to Visit 2.
* Participated in any other studies involving investigational or marketed products within 30 days prior to entry into the study or participated in studies which involved norastemizole, or monoclonal anti-immunoglobulin E (IgE) antibody within 90 days prior to entry into the study.
* Donated blood or blood products for transfusion within 30 days prior to initiation of treatment with study drug and at any time during the study.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 683 (Actual)
Dates: Start 2001-03; Primary Completion 2001-07 (Actual); Study Completion 2001-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline to the Overall endpoint in the subject 24-hour reflective total symptom severity complex (TSSC) score | 2 weeks

SECONDARY OUTCOMES:
Change from baseline to the Overall endpoint in the subject 24-hour reflective TSSC, with and without stuffy nose score | 2 weeks
  Subject rated reflective TSSC on 5-point scale
Change from baseline to the Overall endpoint in the individual rhinoconjunctivitis symptoms (reflective and instantaneous) | 2 weeks
  Subject rated individual symptom severity on 5-point scale (reflective and instantaneous)
Investigator evaluation of rhinoconjunctivitis symptoms | 2 weeks
  Change from baseline to all secondary time points (Week 1 [average of TSSC scores during Week 1 of double-blind treatment], Week 2 [average of TSSC scores during Week 2 of double-blind treatment], and Endpoint [last available post-baseline TSSC score]) in subject 24-hour reflective TSSC.
Parent/legal guardian evaluation of subject's rhinoconjunctivitis symptoms | 2 weeks
  Change from baseline to all secondary time points (Week 1 [average of TSSC scores during Week 1 of double-blind treatment], Week 2 [average of TSSC scores during Week 2 of double-blind treatment], and Endpoint [last available post-baseline TSSC score]) in subject 24-hour reflective TSSC.
Investigator Global Evaluations of Efficacy at Visit 4/early termination | 2 weeks
  Investigator assess the therapeutic regimen's effect on 7-point scale
Subject/Parent/Legal Guardian Global Evaluations at Visit 4/early termination | 2 weeks
  Subject/Parent/Legal Guardian provided global evaluation of treatment on a 5-point scale
Parent/Legal Guardian Overall Personal Satisfaction Assessment at Visit 4/early termination | 2 weeks
  Parent/Legal Guardian provided appraisal of overall personal satisfaction with treatment on a 5-point scale
Parental Burden Questionnaire | 2 weeks
  At Visits 2, 3, and 4/early termination, the parent/legal guardian assessed the social and emotional impact of caring for a child with SAR on a 5-point scale

CONTACTS AND LOCATIONS:
Overall Officials: Dial Hewlett, MD, Study Director — Medical Director; Pfizer, Inc.

IPD SHARING:
Plan to Share IPD: Yes